CLINICAL TRIAL: NCT03682146
Title: A Multicenter Randomized Study to Investigate the Outcomes of Laparoscopic and Robotic-assisted Radical Prostatectomy
Brief Title: Laparoscopic vs Robotic-Assisted Radical Prostatectomy
Acronym: LAP-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Klinikum Dortmund (Unknown); University Hospital Heidelberg (Other); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Jens-Uwe Stolzenburg, Prof., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LAP-01; 110462 (Other Grant/Funding Number: Deutsche Krebshilfe)
Record Dates: First submitted 2015-05-15; First posted 2018-09-24 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: DaVinci; Robotic-Assisted; Prostatectomy; Laparoscopy; Continence
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prostatectomy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were blinded with respect to the surgical method until the end of the 3-month evaluation and extraction of the primary study outcome.
Oversight: Data Monitoring Committee: No

ARMS (2):
- RARP (Other): robot-assisted laparoscopic prostatectomy
  Interventions: Procedure: Prostatectomy
- LRP (Other): conventional laparoscopic radical prostatectomy
  Interventions: Procedure: Prostatectomy

INTERVENTIONS:
Procedure: Prostatectomy — Comparison of robotic-assisted and conventional laparoscopic radical prostatectomy
  Other Names: robotic-assisted laparoscopic radical prostatectomy; conventional laparoscopic radical prostatectomy

SUMMARY:
This randomized trial was designed to address the lack of high-quality literature comparing robotic-assisted (RARP) and laparoscopic (LRP) radical prostatectomy (RP).

Purpose: The LAP-01 trial compares outcomes between RARP and LRP.

DETAILED DESCRIPTION:
LAP-01 is the first multicenter, prospective randomized, patient-blinded controlled trial comparing robotic-assisted and conventional laparoscopic radical prostatectomy.

The investigation include an extensive evaluation of clinical, oncological, functional and quality of life related data by means of validated patient-reported outcome measures.

The primary outcome is the assessment of time to continence restoration at 3 months. This is evaluated by an assessment of a pad diary completed daily by each patient from the time of catheter removal until restoration of continence. Secondary endpoints include continence and erectile function, as well as quality of life (EORTC-QLQ-C30, EORTC-QLQ-PR25), patient satisfaction and Hospital Anxiety and Depression Scale (HADS) at 1, 3, 6 and 12 months after surgery in addition to oncological outcomes up to 3 years follow-up.

With 782 enrolled patients it is the largest trial carried out till date on this topic.

ELIGIBILITY:
Inclusion criteria

* Histological verified prostate carcinoma (first diagnosis)
* Indication for primary curative radical prostatectomy
* Age ≤ 75 years
* Patient agrees to randomisation
* Patient is able to fill in the questionnaires on his own
* Patient is willing to provide written informed consent

Exclusion Criteria:

* Insufficient knowledge of German
* Severe cognitive impairment
* Obesity (BMI > 35)
* Current existing severe comorbidities (e.g. liver cirrhosis, second malignancy or relapse of every kind)
* Tumor stage: T4
* Previous malignancy (≤ 3 years before trial participation)
* Neoadjuvant therapy (hormons) within the last 3 months before participation in the trial
* Patient is immuno-compromised
* History of intermittent urinary self-catheterization within the last year
* Psychological disorders (dementia, chronic depression, psychosis)
* Any of the following treatments ≤ 3 months before trial participation: surgery of the sigmoid colon, extended haemorrhoid resection, transurethral needle ablation of the prostate (TUNA), osteosynthesis of the pelvis, salvage prostatectomy
* Patients with chronic urinary infection
* Dialysis patients
* Lacking willingness for data storage and handling in the frame of the trial protocol/aims

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Early Continence | 3 months after removal of the urinary catheter
  The primary outcome is continence recovery at 3 months based on the patient's pad diary; RARP vs. LRP

SECONDARY OUTCOMES:
Continence | 1, 3, 6, 12 months postoperative
  Continence (pad use/day)
Continence | 1, 3, 6, 12 months postoperative
  Continence (ICIQ-SF scores)
Erectile function | 1, 3, 6, 12 months postoperative
  Erectile function questionnaire (including IIEF-5 questionnaire) and information on supportive medication for erection
Health-related quality of life of patients | 1, 3, 6, 12 months postoperative
  Health-related quality of life questionnaire (EORTC QLQ-C30). Raw scores are linearly transformed into a 0-100 point scale. High global health status and functioning scores indicate good QoL, whereas elevated symptom scores represent a high level of symptomology and therefore impaired QoL.
Prostate-specific quality of life of patients | 1, 3, 6, 12 months postoperative
  Prostate-specific quality of life questionnaire (EORTC QLQ-PR25). Raw scores are linearly transformed into a 0-100 point scale. High functioning scores indicate good QoL, whereas elevated symptom scores represent a high level of symptomology and therefore impaired QoL.
Anxiety and depression assessment | 1, 3, 6, 12 months postoperative
  The Hospital Anxiety and Depression Scales (HADS-D)
Patient satisfaction | 1, 3, 6, 12 months postoperative
  Patient satisfaction is measured on a 5-point scale ranging from highly dissatisfied to highly satisfied. Additionally, patients are asked if they would in hindsight make a decision for or against the surgery and if they would advise a friend to undergo surgery under the same circumstances.
PSA (prostate-specific antigen) | 1, 3, 6, 12, 24, 36 months postoperative
  PSA (prostate-specific antigen)
Rate of relapse and metastases | 1, 3, 6, 12, 24, 36 months postoperative
  Relapse and metastases
Rate of patients with further anti-cancer therapy | 1, 3, 6, 12, 24, 36 months postoperative
  Further anti-cancer therapy
Time of surgery | measured as time from starting the surgical procedure in the DaVinci console to ending the procedure in the console
  time of surgery
Tumor Resection | during surgery
  Tumor Resection
Intra-operative parameters | during surgery
  Rate of Complications

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Uwe Stolzenburg, Prof., Principal Investigator — Leipzig University, Department of Urology
Locations (4):
- Germany (4):
  - Klinikum Dortmund, Dortmund
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - University Hospital Heidelberg, Heidelberg
  - University of Leipzig, Leipzig

REFERENCES:
- [Derived] Holze S, Kuntze AS, Mende M, Neuhaus P, Truss MC, Do HM, Dietel A, Franz T, Stolzenburg JU. Assessment of different continence definitions in the context of the randomized multicenter prospective LAP-01 trial-Does the best definition change over time? Eur J Med Res. 2024 Jan 18;29(1):58. doi: 10.1186/s40001-024-01662-5. PMID 38238789
- [Derived] Holze S, Braunlich M, Mende M, Arthanareeswaran VK, Neuhaus P, Truss MC, Do HM, Dietel A, Franz T, Teber D, Heilsberg AK, Hohenfellner M, Rabenalt R, Albers P, Stolzenburg JU. Age-stratified outcomes after radical prostatectomy in a randomized setting (LAP-01): do younger patients have more to lose? World J Urol. 2022 May;40(5):1151-1158. doi: 10.1007/s00345-022-03945-0. Epub 2022 Feb 6. PMID 35124734
- [Derived] Stolzenburg JU, Holze S, Neuhaus P, Kyriazis I, Do HM, Dietel A, Truss MC, Grzella CI, Teber D, Hohenfellner M, Rabenalt R, Albers P, Mende M. Robotic-assisted Versus Laparoscopic Surgery: Outcomes from the First Multicentre, Randomised, Patient-blinded Controlled Trial in Radical Prostatectomy (LAP-01). Eur Urol. 2021 Jun;79(6):750-759. doi: 10.1016/j.eururo.2021.01.030. Epub 2021 Feb 9. PMID 33573861

DOCUMENTS (1):
  • Study Protocol (2014-02-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT03682146/Prot_000.pdf